CLINICAL TRIAL: NCT01707030
Title: Web-based Intervention to Reduce Alcohol Use in Veterans With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 12-009
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C; Alcohol Abuse
Keywords: clinical trial; veteran; substance use disorder
MeSH Terms: conditions — Hepatitis C; Alcoholism; Substance-Related Disorders | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAI Arm (Experimental): Receiving a web-based brief intervention for alcohol problems
  Interventions: Other: Web-Based Brief Alcohol Intervention; Other: Usual Care
- Usual Care (Active Comparator): In usual care, Hepatitis C clinic staff will sometimes discuss alcohol use with patients, and this will be the experience of some of the controls
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Web-Based Brief Alcohol Intervention — Participants report their alcohol use and problems on line and receive feedback comparing them to national norms.
  Arms: BAI Arm
Other: Usual Care — All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.

SUMMARY:
Many people who are infected with Hepatitis C misuse alcohol, which is even more dangerous for them than it is for a non-infected person. In this VA study, such individuals will be screened and given feedback on their drinking using an Internet-based program which has been shown to reduce drinking in other populations. The research team will evaluate whether the program helps Veterans drink less over time and thereby improve their health.

DETAILED DESCRIPTION:
As many as 80% of Veterans with the hepatitis C virus (HCV) engage in harmful drinking. This is a major health challenge given that even light and moderate alcohol consumption can worsen the course and consequences of HCV and can be a barrier to receiving antiviral therapy. In response, the VA Uniform Mental Health Services Package has made it a priority that HCV and other ambulatory clinics provide evidence-based mental health services to all Veterans engaging in harmful drinking within two week (but preferably the same day as the clinic visit). The investigators' CREATE partners, the VA Office of Mental Health Services, VA Operations (10N), and the VA Office of Public Health, are strongly committed to achieving this standard throughout the Veterans Health Administration (VHA). However, the cost and organizational challenges to meeting this mandate in HCV clinics are enormous, but may be surmountable through the use of self-directed technology that minimizes demands on scarce staff time.

The primary objective of this study is to implement and evaluate a web-based brief alcohol intervention (BAI) for treating Veterans with HCV and seeking care at two VA HCV clinics - Veterans Affairs Palo Alto Health Care System (VAPAHCS) and San Francisco Veterans Affairs Medical Center (SFVAMC). This study will have three aims: First (Aim 1), the investigators plan to assess patient, provider, and system factors that may impact the initial adoption of this intervention in two VA HCV clinics. These data will result in the development of a protocol for the initial implementation of the web-based BAI at the investigators' two study sites. A secondary aim will involve obtaining patient and provider feedback on an existing web-based BAI (see www.bmi-aft.org, VA Intranet Only) to help inform its redesign for use with this population. Second (Aim 2), the investigators will implement and examine the effectiveness of a web-based BAI in two HCV clinics to reduce alcohol consumption in Veterans with HCV at three- and six-months post-treatment. Third (Aim 3), the investigators will conduct a budget impact analysis to estimate the short-term costs (1-3 years) of adoption and diffusion of the web-based BAI and the trajectory of health care spending for study participants.

This mixed-methods study will utilize qualitative and quantitative methods to achieve its three primary aims. To address aim 1, qualitative interviews will be used to collect data that will inform the initial implementation and re-versioning of a web-based BAI for use in two HCV clinics located at the Palo Alto and San Francisco. To address aim 2, the investigators will use a randomized, hybrid (type 1) design with patient level clinical outcome data and formative evaluation data collected to examine the effectiveness of the web-based BAI. "Hybrid" designs also integrate formative evaluation into experimental designs to identify factors that impact the effectiveness of implementation efforts. Formative evaluation (e.g., site visits, clinic observation, and interviews with staff and patients) will be used to improve the adoption of the web-based BAI at both sites and to provide evidence-based guidance to the investigators' CREATE operational partners for nationwide implementation. To address aim 3, the investigators will conduct a budget impact analysis to estimate the short-term costs (1-3 years) of adoption and diffusion of the web-based BAI and the trajectory of health care spending for study participants. The investigators plan to collect several types of utilization data, including outpatient, inpatient, and pharmacy utilization, and calculate total dollars.

ELIGIBILITY:
Inclusion Criteria:

* Must be a US military veteran.
* Over the age of 17 with liver disease.
* Must be receiving care at a VA liver clinic.

Exclusion Criteria:

* Those with no current or historical use of alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith N. Humphreys, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; Michael A Cucciare, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timko C, Schultz NR, Cucciare MA, Vittorio L, Garrison-Diehn C. Retention in medication-assisted treatment for opiate dependence: A systematic review. J Addict Dis. 2016;35(1):22-35. doi: 10.1080/10550887.2016.1100960. Epub 2015 Oct 14. PMID 26467975
- [Result] Cucciare MA, Timko C. Bridging the gap between medical settings and specialty addiction treatment. Addiction. 2015 Sep;110(9):1417-9. doi: 10.1111/add.12977. No abstract available. PMID 26223170
- [Result] Cucciare MA, Cheung RC, Rongey C. Treating substance use disorders in patients with hepatitis C. Addiction. 2015 Jul;110(7):1057-9. doi: 10.1111/add.12893. Epub 2015 Mar 27. No abstract available. PMID 25816843
- [Result] Timko C, Kong C, Vittorio L, Cucciare MA. Screening and brief intervention for unhealthy substance use in patients with chronic medical conditions: a systematic review. J Clin Nurs. 2016 Nov;25(21-22):3131-3143. doi: 10.1111/jocn.13244. Epub 2016 May 3. PMID 27140392
- [Result] Cucciare MA, Jamison AL, Combs AS, Joshi G, Cheung RC, Rongey C, Huggins J, Humphreys K. Adapting a computer-delivered brief alcohol intervention for veterans with Hepatitis C. Inform Health Soc Care. 2017 Dec;42(4):378-392. doi: 10.1080/17538157.2016.1255628. Epub 2017 Jan 9. PMID 28068154
- [Result] Cucciare MA, Combs AS, Joshi G, Han X, Humphreys K. Computer-delivered brief alcohol intervention for patients with liver disease: a randomized controlled trial. Addiction. 2021 May;116(5):1076-1087. doi: 10.1111/add.15263. Epub 2020 Oct 6. PMID 32924207

RESULTS

PARTICIPANT FLOW:
Groups:
- Web-Based BAI Arm: Receiving a web-based brief intervention for alcohol problems
  Web-Based Brief Alcohol Intervention: Participants report their alcohol use and problems on line and receive feedback comparing them to national norms.
- Usual Care Arm: In usual care, Hepatitis C clinic staff will sometimes discuss alcohol use with patients, and this will be the experience of some of the controls
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
Period: Overall Study
Arm/Group | Web-Based BAI Arm | Usual Care Arm
Started | 67 | 71
Completed | 56 | 54
Not Completed | 11 | 17
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Computer-Based Brief Alcohol Intervention: Receiving a web-based brief intervention for alcohol problems
  Web-Based Brief Alcohol Intervention: Participants report their alcohol use and problems on line and receive feedback comparing them to national norms.
  Intervention participants will also receive usual care.
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
- Control: Treatment as Usual: In usual care, Hepatitis C clinic staff will sometimes discuss alcohol use with patients, and this will be the experience of some of the controls
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
- Total: Total of all reporting groups
Arm/Group | Intervention: Computer-Based Brief Alcohol Intervention | Control: Treatment as Usual | Total
Number analyzed (Participants) | 67 | 71 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 82
  >=65 years | 25 | 31 | 56
Age, Continuous [Median (Standard Deviation); unit: years] | 64 (8.682) | 63 (7.212) | 63.5 (8.023)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 62 | 71 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian and/or Pacific Islander | 2 | 1 | 3
  Race/Ethnicity: Black/African Amerian | 21 | 20 | 41
  Race/Ethnicity: White/Caucasion, not of Hispanic origin | 25 | 28 | 53
  Race/Ethnicity: Hispanic | 9 | 15 | 24
  Race/Ethnicity: Other | 6 | 6 | 12
  Race/Ethnicity: Declined to State/Unknown | 1 | 1 | 2
  Race/Ethnicity: American Indian or Alaskan Native | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 71 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change in Days of Unhealthy Alcohol Consumption
Description: The number of days on which alcohol was consumed beyond recommended levels in the last 30 days.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants were able to complete all follow-ups in their entirety. We used an analytical approach that used all available data for the participants for the regression analysis even if participants did not complete all the follow-ups.
Measure: Mean (Standard Deviation); unit: Unhealthy drinking days in last 30
Arm/Group | BAI Arm | Usual Care
Number analyzed (Participants) | 67 | 70
Unhealthy drinking days in last 30
  Baseline Days of Unhealthy Alcohol Consumption | 5.46 (9.24) | 7.16 (10.66)
  3-mo Days of Unhealthy Alcohol Consumption: number analyzed (Participants) | 61 | 57
  3-mo Days of Unhealthy Alcohol Consumption | 2.72 (6.69) | 5.56 (10.68)
  6-mo Days of Unhealthy Alcohol Consumption: number analyzed (Participants) | 56 | 54
  6-mo Days of Unhealthy Alcohol Consumption | 2.29 (6.37) | 4.78 (9.91)

2. Primary Outcome: Change in Drinking Days
Description: The number of days on which alcohol was consumed at any level in the last 30 days.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants were able to complete all questions and/or follow-ups in their entirety. We used an analytical approach that used all available data for the participants for the regression analysis even if participants did not complete all the follow-ups.
Measure: Mean (Standard Deviation); unit: Number of drinking days in last 30
Groups:
- Intervention: Web Based BAI: Receiving a web-based brief intervention for alcohol problems
  Web-Based Brief Alcohol Intervention: Participants report their alcohol use and problems on line and receive feedback comparing them to national norms.
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
- Control: Usual Care: In usual care, Hepatitis C clinic staff will sometimes discuss alcohol use with patients, and this will be the experience of some of the controls
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
Arm/Group | Intervention: Web Based BAI | Control: Usual Care
Number analyzed (Participants) | 67 | 71
Number of drinking days in last 30
  Baseline drinking days: number analyzed (Participants) | 67 | 70
  Baseline drinking days | 9.39 (10.44) | 12.41 (11.47)
  3-mo drinking days: number analyzed (Participants) | 61 | 57
  3-mo drinking days | 5.20 (8.09) | 7.77 (10.78)
  6-mo drinking days: number analyzed (Participants) | 56 | 54
  6-mo drinking days | 4.61 (7.66) | 8.26 (10.67)

3. Secondary Outcome: Change in Drinks Per Drinking Day
Description: The number of standard drinks (0.5 ounce ethanol equivalent) consumed on those days that an individual drank in the last 30 days.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Drinks per Drinking Day
Arm/Group | Intervention: Web Based BAI | Control: Usual Care
Number analyzed (Participants) | 67 | 71
Drinks per Drinking Day
  Baseline Drinks per Drinking Day: number analyzed (Participants) | 67 | 70
  Baseline Drinks per Drinking Day | 3.57 (3.90) | 3.72 (3.69)
  3-mo Drinks per Drinking Day: number analyzed (Participants) | 61 | 57
  3-mo Drinks per Drinking Day | 2.29 (2.47) | 2.17 (2.17)
  6-mo Drinks per Drinking Day: number analyzed (Participants) | 56 | 54
  6-mo Drinks per Drinking Day | 1.98 (2.85) | 1.87 (1.90)

4. Secondary Outcome: Change in Symptoms of Psychological Distress (PHQ-9)
Description: Symptoms of psychological distress will be measured using the Patient Health Questionnaire (PHQ-9). The PHQ-9 provides an assessment of depression severity. The minimum value is 0 and the maximum value is 27. Lower scores are better. The reliability, validity, and clinical utility of the PHQ-9 instrument are well-established.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Web Based BAI | Control: Usual Care
Number analyzed (Participants) | 67 | 71
score on a scale
  Baseline PHQ-9 | 6.00 (5.70) | 6.68 (5.67)
  3-mo PHQ-9: number analyzed (Participants) | 61 | 57
  3-mo PHQ-9 | 6.03 (5.65) | 6.91 (6.86)
  6-mo PHQ-9: number analyzed (Participants) | 56 | 54
  6-mo PHQ-9 | 5.57 (5.07) | 7.44 (7.48)

5. Secondary Outcome: Change in SF-12 Physical Health Composite
Description: The Short Form-12 (SF-12) is a 12-item health survey based on the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) designed to assess two component health status summary scales (physical and mental component summaries) in the general U.S. population . The SF-12 has demonstrated good internal consistency reliability and construct validity. This reflects the physical health component of the SF-12. Scores range from 0-100 and higher scores are better.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Web Based BAI | Control: Usual Care
Number analyzed (Participants) | 67 | 71
score on a scale
  Baseline SF-12 Health: number analyzed (Participants) | 67 | 70
  Baseline SF-12 Health | 40.43 (12.20) | 40.49 (11.43)
  3mo SF-12 Health: number analyzed (Participants) | 60 | 55
  3mo SF-12 Health | 39.92 (12.25) | 41.59 (12.30)
  6mo SF-12 Health: number analyzed (Participants) | 56 | 51
  6mo SF-12 Health | 42.21 (10.43) | 40.75 (12.45)

6. Secondary Outcome: Change in Additional Care
Description: Total costs in dollars of all VA and non-VA inpatient, outpatient and pharmacy costs.
Time Frame: Baseline and 12 months
Population: These are the same individuals enrolled in the clinical trial from whom the primary outcomes were assessed.
Measure: Mean (Standard Error); unit: US Dollars
Arm/Group | Web-Based BAI Arm | Usual Care Arm
Number analyzed (Participants) | 53 | 54
US Dollars | 42412 (5381) | 51667 (8611)

7. Other Pre Specified Outcome: Change in SF-12 Mental Health Composite
Description: The Short Form-12 (SF-12) is a 12-item health survey based on the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) designed to assess two component health status summary scales (physical and mental component summaries) in the general U.S. population. The SF-12 has demonstrated good internal consistency reliability and construct validity. This reflects the mental health component of the SF-12. Scores range from 0-100 and higher scores are better.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Web Based BAI | Control: Usual Care
Number analyzed (Participants) | 67 | 71
score on a scale
  Baseline SF-12 Mental Health: number analyzed (Participants) | 67 | 70
  Baseline SF-12 Mental Health | 49.10 (12.72) | 48.91 (11.87)
  3mo SF-12 Mental Health: number analyzed (Participants) | 60 | 55
  3mo SF-12 Mental Health | 50.83 (9.94) | 49.25 (11.62)
  6 mo SF-12 Mental Health: number analyzed (Participants) | 56 | 51
  6 mo SF-12 Mental Health | 50.63 (10.59) | 48.51 (12.77)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 4 years.
Groups:
- Intervention: Web-Based BAI Arm: Receiving a web-based brief intervention for alcohol problems
  Web-Based Brief Alcohol Intervention: Participants report their alcohol use and problems on line and receive feedback comparing them to national norms.
- Control: Usual Care Arm: In usual care, Hepatitis C clinic staff will sometimes discuss alcohol use with patients, and this will be the experience of some of the controls
  Usual Care: All patients will be receiving care in a Hepatitis C clinic. In some cases clinicians may counsel them on alcohol problems.
Arm/Group | Intervention: Web-Based BAI Arm | Control: Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 1/67 | 1/71
Serious Adverse Events (participants affected / at risk) | 1/67 | 1/71
Other Adverse Events (participants affected / at risk) | 0/67 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Web-Based BAI Arm (N=67) | Control: Usual Care Arm (N=71)
Death (General disorders) | 1 (1) | 0 (0) — Intervention: Unable to pinpoint cause of death at time of entry as participant had multiple disorders which could have caused death. Control: Renal Disease
Death (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT01707030/Prot_SAP_000.pdf